CLINICAL TRIAL: NCT02915562
Title: Influence of Depressive Mood on Short Term Rehab Outcome at an Acute Geriatrics Unit
Brief Title: Influence of Depressive Mood on Rehab Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Collaborators: Kepler University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PMR-AGR-001
Record Dates: First submitted 2016-04-14; First posted 2016-09-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Depressive Mood
Keywords: rehabilitation; exercise; outcome measurement
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Depressive Group (Active Comparator): GDS 15 (Geriatric Depression Score) ≥5 at baseline
  Interventions: Other: exercise
- Non-depressive Group (Active Comparator): GDS 15 (Geriatric Depression Score) <5 Points at baseline
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise

SUMMARY:
The purpose of this study is to determine the effects of depressive mood on outcomes of an in-house rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* 2-week in-house-rehab at an acute geriatric unit
* ability to take part in assessments
* understanding German language
* Informed Consent

Exclusion Criteria:

* anti-depressive medication shorter than 4 weeks before enrollment
* In-house rehab < 14 days
* advanced stage of dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Physical Performance Test | Change from baseline at day 14 +/-1
de Morton Mobility Index | Change from baseline at day 14 +/-1
  The de Morton Mobility index is a method for measuring changes in mobility and enhancing the continuity of patient care across clinical settings
Performance Orientated Mobility Assessment (POMA) | Change from baseline at day 14 +/-1
  Task-oriented outcome measure that assesses gait and balance ability
Barthel Index | Change from baseline at day 14 +/-1
  The Barthel index is an ordinal scale used to measure performance in activities of daily living
Function Index Physiotherapy | Change from baseline at day 14 +/-1
Function Index Occupational Therapy | Change from baseline at day 14 +/-1
Grip strength measurement | Change from baseline at day 14 +/-1
  measured with JAMAR dynamometer

SECONDARY OUTCOMES:
Charlson Comorbidity Index | Day 1+/-1
  Measure of comorbidity and multimorbidity
Timed Test of Money Counting | Day 1+/-1
Geriatric Depression Scale (GDS-15) | Day 1+/-1 and day 14+/-1

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Hospital, Linz, Austria

IPD SHARING:
Plan to Share IPD: No